CLINICAL TRIAL: NCT04546815
Title: Non-interventional Observational Study of Daptomycin in the Treatment of Gram-positive Bacterial Infections
Brief Title: The Efficacy and Safety of Daptomycin in the Treatment of Gram-positive Bacterial Infection.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: SINGCHN-DAP-IV-2002
Record Dates: First submitted 2020-08-26; First posted 2020-09-14 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Antibiotic
MeSH Terms: interventions — Daptomycin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Gram-positive cocci infection: No intervention. The clinical data of patients (including demographic information, details of anti-infective therapy, imaging and laboratory testings) will be collected and analyzed.
  Interventions: Drug: Daptomycin

INTERVENTIONS:
Drug: Daptomycin — According to the severity of the disease, the site of infection and clinical response, the doctor makes a drug regimen of datoramycin.

SUMMARY:
This study aims to collect and analyze clinical data of daptomycin to explore the efficacy and safety of daptomycin in the treatment of Gram-positive bacterial infections. And optimize the dosing regimen based on these data.

DETAILED DESCRIPTION:
With the gradual increase in the detection rate of drug-resistant bacteria, bloodstream infections, skin and soft tissue infections, infective endocarditis and other infectious diseases caused by MRSA, MRCNS, and VRE have greatly increased patient mortality and medical burden.

Daptomycin has strong anti-bacterial activity and rapid sterilization. It is almost 100% sensitive to common Gram-positive bacteria. Both domestic and foreign guidelines recommend its use for the treatment of infectious diseases such as bacteremia, central venous catheter-related bloodstream infections, infective endocarditis, skin and soft tissue infections, bone and joint infections，and so on. However, there is a lack of actual clinical use of daptomycin in China, as well as efficacy and safety assessments based on real world data.

The purpose of this study is to collect and analyze data on the use of daptomycin in the real world. The clinical cure rate and inefficiency, temperature drop time, 28-day mortality rate are the primary outcome measures, and the overall incidence of adverse events, the results of CPK monitoring and its correlation with dose, renal function, length of hospital stay, and treatment costs are secondary outcome measures to investigate the efficacy and safety of daptomycin in the treatment of gram-positive bacterial infection.

ELIGIBILITY:
Inclusion Criteria:

* 1 years of age or older
* Meet one of the following conditions:

  1. Confirmed Gram-positive cocci (GPC) infection;
  2. Cases evaluated by doctors as suspected gram-positive coccal infection with potentially high benefit from drug use；
  3. Severe infection patients to be combined with empirical treatment of daptomycin.
* The off-label drug use conforms to the relevant administrative regulations of each participating unit.

Exclusion Criteria:

* Allergic to datoramycin;
* Pregnant and lactating women；
* Patients with age < 1 year；
* Participate in other clinical trials；
* Patients with nervous system GPC infection;
* Patients with pulmonary GPC infection.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: The study plans to recruit 2000 patients infected with gram-positive bacteria.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy rate | 1 day of the end of treatment
  Clinical efficacy includes clinical cure and clinical improvement.
Clinical cure rate | 14 days of the end of treatment
  Clinical cure was defined as that after the end of treatment, all the selected symptoms and signs had disappeared or completely returned to normal, and all the non-microbiological indicators, such as imaging and laboratory examination, had returned to normal.
Treatment failure rate | 28 days of the end of treatment
  Treatment failure includes one of the following conditions:
  1. After the end of the treatment, all the symptoms and signs of the patients at the time of inclusion continued or worsened.
  2. Recurrence.
  3. Termination of treatment due to adverse reactions.
Time for body temperature to return to normal. | 14 days of the end of treatment
  During the use of daptomycin, take body temperature records.
28-Day Mortality Rate | 28 days of the end of treatment
  Record the number of deaths 28 days after the end of treatment

SECONDARY OUTCOMES:
Bacteria clearance rate (if available, such as bacteremia) | 1 day of the end of treatment
  Bacterial clearance includes clearance and hypothetical clearance. Bacterial clearance is defined as the specimens from the original infection site after treatment have not cultivated the pathogenic bacteria of the original infection.
  When the patient's symptoms and signs disappear so that cultivable materials cannot be obtained, or the method of obtaining specimens is too invasive for the recovered patient, the bacteriological result is considered to be a hypothetical clearance.
The overall incidence of adverse events | 14 days of the end of treatment
  Adverse events refer to adverse medical events that occur after patients or clinical trial subjects receive a drug, but they do not necessarily have a causal relationship with treatment.
Monitor creatine phosphokinase（CPK） levels | 14 days of the end of treatment
  Record the CPK monitoring results.
hospital stays | 28 days of the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: XiaoJun X Ma, doctor, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The clinical study data of this project were owned by the participating research center. For other researchers who need data, the results of the study can be understood through the literature published later.